CLINICAL TRIAL: NCT03588442
Title: Prospective Surveillance for Very Early Hepatocellular Carcinoma (PRECAR): an Observational Cohort Trial
Brief Title: Prospective Surveillance for Very Early Hepatocellular Carcinoma
Acronym: PRECAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, Lei Chen, PhD, Professor, Eastern Hepatobiliary Surgery Hospital
Other Study IDs: 2018ZX10732202
Record Dates: First submitted 2018-07-01; First posted 2018-07-17 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cirrhosis cohort: Patients with liver cirrhosis.
- HBV infection cohort: Patients with seropositivity of HBsAg.

SUMMARY:
Hepatocellular carcinoma is one the leading cause of increasing cancer-specific mortality worldwide. Early diagnosis of hepatocellular carcinoma provides opportunity for curative therapeutic approaches and relatively favorable prognosis. Herein, we intended to establish a biosignature for early diagnosis of hepatocellular carcinoma and stratification of risk population for intensive follow-up by implementing biannual follow-up investigation and collecting peripheral blood samples for screening.

DETAILED DESCRIPTION:
Patients will be recruited for 1 year and be follow-up for 3 years. Patients will make active hospital visit for collection of blood samples, which will be analyzed to develop a biosignature at the end of the study to detect very early hepatocellular carcinoma and stratify risk population for intensive follow-up.

ELIGIBILITY:
Inclusion Criteria:

-

[1] Cirrhosis cohort

1. Age within 30 to 75 years.
2. Diagnosis of liver cirrhosis within recent 6 months.

<!-- -->

1. Liver biopsy: Metavir score of 4 or Ishak score of 5 to 6.
2. No liver biopsy: Presence of ascites, hepatic encephalopathy, or variceal hemorrhage.
3. Satisfying equal to or more than 2 of below conditions.

   * Imaging studies indicating characteristics of liver cirrhosis: irregular liver surface, liver parenchyma particles or nodules, intraperitoneal collateral circulation, or varicose veins with or without splenomegaly (more than 4 cm or 5 ribs).
   * Platelet count < 200 x 10^9/L.
   * Alanine aminotransferase < 5 folds of normal level and liver hardness > 12 kPa.
   * Gastroesophageal varices from endoscopy or imaging studies.

     [2] HBV infection cohort
     1. Age within 40 to 70 years
     2. Chronic HBV infection (seropositive for HBsAg over 6 months).

        Exclusion Criteria:
        1. Cirrhosis cohort

     (1) Child-Pugh score of C.

     (2) Hereditary metabolic liver diseases.

     (3) Presence of HIV-Ab.

     (4) Previous diagnosis of active pulmonary tuberculosis.

     (5) Diagnosis of malignant tumors before or during hospitalization, including but not limited to hepatocellular carcinoma.

     (6) Patients who had received allogeneic blood transfusion or cell therapy within 1 year.

     (7) Pregnant women.

     [2] HBV infection cohort

     (1) Autoimmune liver diseases.

     (2) Hereditary metabolic liver diseases.

     (3) Other chronic liver diseases, such as flukes.

     (4) Presence of HCV, HDV, HEV, or HIV infection.

     (5) Previous diagnosis of active pulmonary tuberculosis.

     (6) Diagnosis of malignant tumors before or during hospitalization, including but not limited to hepatocellular carcinoma.

     (7) Patients who had received allogeneic blood transfusion or cell therapy within 1 year.

     (8) Pregnant women.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cirrhosis cohort: patients with liver cirrhosis. HBV infection cohort: patients with chronic HBV infection.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2018-07-15 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
Hepatocellular carcinoma | July 2018 to July 2022
  Development of hepatocellular carcinoma
Overall survival | July 2018 to July 2022
  Death
Liver-related disease progression | July 2018 to July 2022
  HBV and cirrhosis progression

SECONDARY OUTCOMES:
Non-hepatocellular carcinoma malignant neoplasm | July 2018 to July 2022
  Development of other primary liver cancer, such as Intrahepatic cholangiocarcinoma.

CONTACTS AND LOCATIONS:
Overall Officials: Hongyang Wang, MD and PhD, Principal Investigator — Eastern Hepatobiliary Surgery Hospital, Second Military Medical University, Shanghai, China; Jinlin Hou, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (13):
- China (13):
  - The First Hospital Affiliated to AMU (Southwest Hospital), Chongqing, Chongqing Municipality
  - Mengchao Hepatobiliary Surgery Hospital of Fujian Medical University, Fuzhou, Fujian
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - Chifeng Municipal Hospital, Chifeng, Inner Mongolia
  - Xuzhou No.1 People's Hospital, Xuzhou, Jiangsu
  - Xuzhou Infectious Disease Hospital, Xuzhou, Jiangsu
  - The First Bethune of Jilin University, Changchun, Jilin
  - The Second Hospital of Shandong University, Jinan, Shandong
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - Shanghai Oriental Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality
  - First Affiliated Hospital, Xinjiang Medical University, Ürümqi, Xinjiang
  - HwaMei Hospital, University of Chinese Academy of Sciences, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xing X, Cai L, Ouyang J, Wang F, Li Z, Liu M, Wang Y, Zhou Y, Hu E, Huang C, Wu L, Liu J, Liu X. Proteomics-driven noninvasive screening of circulating serum protein panels for the early diagnosis of hepatocellular carcinoma. Nat Commun. 2023 Dec 18;14(1):8392. doi: 10.1038/s41467-023-44255-2. PMID 38110372

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/42/NCT03588442/Prot_SAP_000.pdf